CLINICAL TRIAL: NCT02741635
Title: The Evaluation of a Nasal Pillows Mask for the Treatment of Obstructive Sleep Apnea (OSA) in NZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-190
Record Dates: First submitted 2016-04-06; First posted 2016-04-18 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- New Nasal Pillows Mask (Experimental): Participants to use nasal pillows mask one night in lab overnight polysomnography.
  Interventions: Device: New Nasal Pillows Mask

INTERVENTIONS:
Device: New Nasal Pillows Mask — Nasal Pillows mask for the treatment of obstructive sleep apnea (OSA)

SUMMARY:
This investigation is designed to evaluate the performance (leak and comfort) as well as the participant's overall acceptance of the nasal pillows mask amongst Obstructive Sleep Apnea (OSA) participants. Also to assist in the development process it would be beneficial to get feedback from users on certain aspects of the design. The aim of this investigation is to get feedback on the first impressions (look and feel) from users of nasal pillows PAP therapy.

A total number of 15 participants who currently use a nasal pillows mask will be recruited for the trial. Participants from previous NZ trials may be recruited into this trial with their consent. All the participants will be recruited from the Fisher & Paykel Healthcare Database of subjects with OSA (Ethics Reference NTY/08/06/064), Auckland District Health Board (ADHB) and New Zealand Respiratory and Sleep Institute (NZRSI).

Participants will undergo an overnight polysomnography session at the Fisher & Paykel Healthcare sleep lab.

The participant will use the trial device on their usual Continuous or Auto Positive Airway Pressure (CPAP/APAP) setting and device for the duration of the overnight in-lab study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* AHI ≥ 5 on diagnostic night
* Prescribed a CPAP device after successful OSA diagnosis
* Existing nasal pillows mask user

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness.
* Anatomical or physiological conditions making APAP therapy inappropriate
* Commercial drivers who are investigated by New Zealand Transport Agency (NZTA)
* Current diagnosis of CO2 retention
* Pregnant or may think they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavi Ogra, BSc, Principal Investigator — Sponsor Employee
Locations (1):
- Fisher & Paykel Healthcare Ltd, Auckland, East Tamaki, New Zealand

IPD SHARING:
Plan to Share IPD: No
For product development purposes only. Data will be de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Toffee Nasal Pillows Mask: Participants to use nasal pillows mask one night in lab overnight polysomnography.
  New Nasal Pillows Mask: Nasal Pillows mask for the treatment of obstructive sleep apnea (OSA)
Period: Overall Study
Arm/Group | Toffee Nasal Pillows Mask
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Toffee Nasal Pillows Mask: Participants to use nasal pillows mask one night in lab overnight polysomnography.
  Toffee Nasal Pillows Mask: Nasal Pillows mask for the treatment of obstructive sleep apnea (OSA)
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  18+ years of age | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Participants Choose the Toffee Mask Based on First Impressions Over 3 Market Leading Masks
Time Frame: 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 14
Participants | 4

2. Secondary Outcome: Participants Consider the Toffee Mask to be as Comfortable, or Much More Comfortable Than Their Usual Mask
Time Frame: 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 14
Participants | 9

3. Secondary Outcome: Participants Consider the Toffee Mask to be Easier or Much Easier to Fit and Adjust Than Their Current Mask
Time Frame: 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Toffee Nasal Pillows Mask
Number analyzed (Participants) | 14
Participants | 8

ADVERSE EVENTS:
Arm/Group | Toffee Nasal Pillows Mask
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No